CLINICAL TRIAL: NCT06447740
Title: Fractional Flow Reserve-guided Percutaneous Renal Artery Stenting Plus Optimal Medical Therapy Versus Optimal Medical Therapy Alone In Atherosclerosis Renal-vascular Hypertension Patients: a Multicenter Randomized Trial
Brief Title: Fractional Flow Reserve-guided Stenting Versus Medical Therapy in Atherosclerosis Renal Artery Stenosis
Acronym: FAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024研210-002
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Renal Artery Stenosis Atherosclerotic; Secondary Hypertension Renal Arterial
MeSH Terms: interventions — Dopamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stenting plus OMT with FFR <0.80 (Experimental)
  Interventions: Drug: Dopamine; Diagnostic Test: Fractional Flow Reserve, Renal; Device: Renal artery stenting
- OMT alone with FFR < 0.80 (Placebo Comparator)
  Interventions: Drug: Dopamine; Diagnostic Test: Fractional Flow Reserve, Renal
- OMT alone with FFR ≥0.80 (Other)
  Interventions: Drug: Dopamine; Diagnostic Test: Fractional Flow Reserve, Renal

INTERVENTIONS:
Drug: Dopamine — A bolus dose of 50μg/kg dopamine via renal artery to induce hyperemic status
Diagnostic Test: Fractional Flow Reserve, Renal — Renal FFR will be measured based on SOP
Device: Renal artery stenting — Renal artery stenting will be implanted based on the protocol
  Arms: Stenting plus OMT with FFR <0.80

SUMMARY:
Although randomized trials have demonstrated there is no benefit of renal-artery stenting in addition to medical therapy for patients with atherosclerosis renal artery stenosis, many patients indeed gained benefit in daily practices after stenting, such as reduction in blood pressure and recovery in renal functions. One important gap is that there is no universal standard to determine whether to stent in these patients. Fraction Flow Reserve (FFR) has been studied for many year in chronic coronary heart disease and FFR-guided revascularization strategy is known to be better than both angiography-guided revascularization and medication alone. Based on the primary finding of FAIR-pilot study (NCT05732077), FFR-guided renal artery stenting is practical.

The overall purpose of the FAIR trial is to compare the clinical outcomes and safety of FFR-guided stenting plus optimal medical treatment (OMT) versus OMT alone in patients with renal-vascular hypertensive patients.

With the 'all comers' design, participants met the inclusive/exclusive criteria will be enrolled, and hyperemic FFR induced by dopamine will be measured in all participants. If FFR is ≥0.80, patients will be treated with OMT alone and follow up. If FFR is <0.80, participants will be randomized to stenting in the renal artery plus OMT or OMT alone on a 1:1 ratio. The blood pressure and anti-hypertensive medications will be compared before and 3 months after the procedure based on ambulatory blood pressure monitoring, all participants will be followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* With recorded hypertension, AND the blood pressure is not controlled (daytime mean SBP ≥135 mmHg and/or DBP ≥85 mmHg based on ABPM) on 2 or more classes of anti-hypertensive drugs;
* Evidence of renal artery stenosis and undergoing renal artery angiography;
* Able to follow the study protocol and provide informed consent;
* Renal artery angiography shows at least 1 main artery with stenosis of 50%-90%, AND the diameter is ≥ 4.0mm.

Exclusion Criteria:

* SBP ≥200mmHg and/or DBP ≥120mmHg at the day or randomization;
* Fibromuscular dysplasia or other non-atherosclerotic renal artery stenosis;
* Pregnancy or unknown pregnancy status in female of childbearing potential;
* Participation in any drug or device trial during the study period;
* Any stroke/TIA, OR with ≥70% stenosis of carotid artery;
* Any major surgery, myocardial infarction or interventional therapy 30 days prior to study entry;
* LVEF <30%;
* Comorbidity condition causing life expectancy ≤1 year;
* Allergy to contrast or any of the following: aspirin, clopidogrel;
* Previous kidney transplant;
* Previous renal artery bypass surgery or stent intervention;
* Kidney size less than 8 cm measured by ultrasound;
* Local lab serum Cr >3.0 mg/dl (265.2μmol/l) on the day of randomization;
* Reference vessel size <4 mm or >8 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Change in daytime mean systolic blood pressure as measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM) | From baseline to 3 months post-procedure
Change in the composite index of antihypertensive drugs | From baseline to 3 months post-procedure
  Change in the composite index of antihypertensive drugs. Drug Composite Index = Weight (number of classes of antihypertensive drugs) × (sum of doses)

SECONDARY OUTCOMES:
Change in systolic blood pressure as measured by 24-hour ABPM | From baseline to 3 months post-procedure
Change in diastolic blood pressure as measured by 24-hour ABPM | From baseline to 3 months post-procedure
Change in home blood pressure | From baseline to 3 months post-procedure
Change in office blood pressure | From baseline to 3 months post-procedure
Change in the composite index of antihypertensive drugs to reach target blood pressure | From baseline to 1 year post-procedure
  Change in the composite index of antihypertensive drugs to reach target blood pressure. Drug Composite Index = Weight (number of classes of antihypertensive drugs) × (sum of doses)
Change in ABPM | From baseline to 6 months, 1 year post-procedure
All-cause death | From baseline to 1 year post-procedure
Cardiac death | From baseline to 1 year post-procedure
Acute myocardial infarction incidence | From baseline to 1 year post-procedure
  Based on universal definition of acute myocardial infarction
Non-fatal stroke incidence | From baseline to 1 year post-procedure
  Based on medical records under outcome committee's judge
Rehospitalization due to heart failure incidence | From baseline to 1 year post-procedure
  Based on medical records under outcome committee's judge
Change in serum creatinine or dialysis | From baseline to 1 year post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China